CLINICAL TRIAL: NCT05263128
Title: Validity Study of the Turkish Version of the Hand20 Questionnaire With Carpal Tunnel Syndrome
Brief Title: Turkish Version of the Hand20 Questionnaire With Carpal Tunnel Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: The research was left unfinished and was not continued.
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Neslihan Torun, Investigator, Hasan Kalyoncu University
Other Study IDs: Hasan Kalyoncu Universty
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boston carpal tunnel syndrome questionnaire
  Interventions: Other: Investigation of the validity of the Hand-20 Questionnaire in individuals with carpal tunnel syndrome
- Hand-20 questionnaire
  Interventions: Other: Investigation of the validity of the Hand-20 Questionnaire in individuals with carpal tunnel syndrome

INTERVENTIONS:
Other: Investigation of the validity of the Hand-20 Questionnaire in individuals with carpal tunnel syndrome — To investigate the validity and reliability of the Hand-20 questionnaire used in individuals with upper extremity disease by comparing it with the Boston carpal tunnel syndrome questionnaire in individuals with carpal tunnel syndrome in Turkey

SUMMARY:
The questionnaire will be investigated by administering the Hand-20 questionnaire and the Boston Carpal Tunnel Syndrome Questionnaire to patients with carpal tunnel syndrome, one week apart.

DETAILED DESCRIPTION:
Questionnaires, which are used to express the perception of difficulty and hand functionality during daily living activities of individuals with carpal tunnel syndrome, and most importantly, which are easy to administer, should be preferred in order to plan a patient-specific treatment program with these results. Self-administered questionnaires showing the physical dimension of recovery are effective and sensitive to change.

Hand20 is a short, easy-to-understand and visual questionnaire used to evaluate disorders caused by upper extremity pathologies, developed by Suzuki et al. in 2010 and proven to be valid in upper extremity diseases by Töre et al. In this questionnaire consisting of 20 questions, the answer to each question is graded between 0 and 10 (0: No restrictions, 10: Impossible). The best score is 0, the worst score is 100.

Boston carpal tunnel syndrome questionnaire (BKTSA) will be used to evaluate the functionality level and symptom severity of the patients. In this questionnaire, which consists of 2 parts: symptom severity and functional capacity, a separate average score will be calculated for each part by dividing the total score obtained by the number of questions. An increased score indicates decreased functional capacity and increased symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25-60 years
* Patients diagnosed with carpal tunnel
* Patients who volunteered for treatment

Exclusion Criteria:

* Patients who do not agree to volunteer
* Patients who have undergone surgery from the wrist region

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Individuals diagnosed with carpal tunnel syndrome
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Investigation of the Validity of the Hand-20 Questionnaire in Individuals with Carpal Tunnel Syndrome | 1 week apart

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University

IPD SHARING:
Plan to Share IPD: No